CLINICAL TRIAL: NCT03801915
Title: Perioperative MVT-5873, a Fully Human Monoclonal Antibody Against a CA 19-9 Epitope, for Operable CA 19-9 Producing Pancreatic Cancers, Cholangiocarcinomas, and Metastatic Colorectal Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jonathan Hernandez, M.D., Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 190039; 19-C-0039
Record Dates: First submitted 2019-01-11; First posted 2019-01-14 (Actual); Results first posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-02

CONDITIONS: Colon Cancer; Pancreatic Cancer; Cholangiocarcinoma; Metastatic Colon Carcinoma; Liver Metastasis
Keywords: Well Tolerated Agent; Pancreas and Liver Resections; Recurrence-Free Survival
MeSH Terms: conditions — Colonic Neoplasms; Pancreatic Neoplasms; Cholangiocarcinoma | interventions — Pancreatectomy; Hepatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 - Pre-operative Escalation Doses of MVT-5873 (HuMab-5B1) (Experimental): Pre-operative escalation doses of MVT-5873, pancreatectomy or hepatectomy and post-operative MVT-5873 treatment
  Interventions: Drug: MVT-5873; Procedure: pancreatectomy or hepatectomy
- Cohort 2 - Pre-operative Recommended Dose (RD) of MVT-5873 (HuMab-5B1) (Experimental): Pre-operative RD of MVT-5873, pancreatectomy or hepatectomy and post-operative MVT-5873 treatment
  Interventions: Drug: MVT-5873; Procedure: pancreatectomy or hepatectomy

INTERVENTIONS:
Drug: MVT-5873 — 1 mg/kg or 3 mg/kg for pre-operative dose, 1 mg/kg during post-operative period
  Other Names: HuMab-5B1
Procedure: pancreatectomy or hepatectomy — Pancreatectomy or hepatectomy

SUMMARY:
Background:

Gastrointestinal tumors have a molecule called carbohydrate antigen 19-9 (CA19-9) in the tumors and blood. The agent MVT-5873 was designed to block this molecule. Researchers want to test how safe it is to give this agent to people before and after surgery to remove a tumor. They want to learn the highest dose tolerated. They want to see if getting the agent at surgery helps slow down the disease.

Objective:

To test the safety of giving MVT-5873 at surgery to remove cancer and see if it slows the progression of the disease.

Eligibility:

Adults at least 18 years old with certain cancers and certain blood CA19-9 levels

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Blood and heart tests
* Scans
* Review of normal activities
* Review of tumor sample
* Pregnancy test

A few days before surgery, participants will get a dose of the study agent. They will get it through a small plastic tube in a vein over about 2 hours.

Participants will sign a separate consent and have the surgery. A sample of the tumor and normal liver will be removed for research.

For 1-2 weeks after surgery, participants will recover in intensive care then regular care at the hospital. They will be monitored and treated throughout the stay.

After leaving the hospital, participants will get the study agent every week for 1 month. Then they will get it every other week for 2 months. They will repeat screening tests at study visits and at a follow-up visit. That will be about 5 weeks after the last dose.

DETAILED DESCRIPTION:
Background:

* Resections to remove tumors in the liver, bile ducts and pancreas are rarely curative, and patients frequently succumb to disease recurrence in the ensuing months to year(s) after the operation.
* Standard adjuvant therapies, which typically begin 6-12 weeks after surgery, offer little demonstrable decreases in the rates of tumor recurrence.
* The concept and implementation of immediate perioperative therapy has not been evaluated given the serious concerns related to healing and recovery with standard cytotoxic chemotherapy and newer targeted agents.
* A significant percentage of metastatic colorectal cancers, and primary tumors of the pancreas and bile ducts express Sialyl Lewis, an epitope on the well-established tumor marker, Carbohydrate antigen 19-9 (CA19-9).
* MVT-5873, a fully human antibody against Sialyl Lewis, has displayed antibody-dependent cell-mediated cytotoxicity (ADCC) and complement dependent cytotoxicity (CDC) in vitro, potentiated chemotherapeutic efficacy in mouse models and demonstrated efficacy in Phase 1 trials of patients with advanced inoperable Hepato-pancreato-biliary (HPB) cancers.
* MVT-5873 is well tolerated as a single agent; moderate elevations in aspartate aminotransferase (AST)/alanine aminotransferase (ALT) appear to be dose-limiting.
* Patients with resectable Sialyl Lewis-expressing cancers represent an ideal population to explore the use of perioperative MVT-5873 given moderate level of CA 19-9 elevations, and the potential for extension of recurrence-free survival.

Objectives:

* Document the safety of perioperative MVT-5873 in patients undergoing pancreas and liver resections.
* Determine if perioperative MVT-5873 can decrease 1-year recurrence rates for patients with operable CA 19-9-producing cancers.

Eligibility:

* Histologically or cytologically confirmed adenocarcinoma of the

  * Colon (metastatic to liver)
  * Pancreas
  * Bile Ducts (Cholangiocarcinoma)
* Serum CA19-9 levels greater than the upper limit of normal, but less than 2500.
* Disease amenable to complete surgical extirpation.

Design:

-Pre-operative one-time treatment with MVT-5873, resection to remove all demonstrable disease in the liver, bile ducts and pancreas, and continuing MVT-5873 mono-therapy until off treatment criteria are met.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects must have histologically or cytologically confirmed diagnoses of adenocarcinoma in one of the following scenarios:

  * Primary tumors of the pancreas
  * Primary tumors of the bile duct and ampulla
  * Metastatic colorectal cancers to the liver
* Subjects must have disease resectable with a standard pancreatectomy (pancreaticoduodenectomy or distal pancreatectomy) or liver resection.
* Subjects may have received prior therapy, including neoadjuvant regimens.
* Subjects must have serum Carbohydrate antigen 19-9 (CA 19-9) elevations greater than the upper limit of normal but less than 2500 U/mL.
* Age greater than or equal to 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1
* Subjects must have adequate organ and marrow function as defined below:

  * leukocytes >3,000/mcL
  * absolute neutrophil count >1,500/mcL
  * platelets >90,000/mcL
* For subjects with Periampullary cancers that require a pancreaticoduodenectomy for complete tumor extirpation:

  * total bilirubin <10 upper limit of normal (ULN)*
  * Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamate-pyruvate transaminase (SGPT) <5 X institutional upper limit of normal
  * creatinine <1.5X institutional upper limit of normal

    * Subjects with periampullary cancers typically present with biliary obstruction resulting in significant abnormalities in liver function tests that do not reflect liver dysfunction. These values normalize after tumor removal. They can be normalized pre-operatively with biliary stenting, but several large studies have demonstrated an increase in infectious complications with drainage. As such, a practice standard has been to avoid stenting until bilirubin level rises above 10 X ULN.
* For subjects with liver tumors (cholangiocarcinoma or metastatic colorectal cancer) requiring a hepatectomy for complete tumor extirpation:

  * total bilirubin <2.5 X institutional upper limit of normal*
  * AST(SGOT)/ALT(SGPT) <5 X institutional upper limit of normal*
  * creatinine <1.5X institutional upper limit of normal

    * Liver abnormalities in this range are consistent with parenchymal destruction from the tumor.
* For subjects with pancreas tumors that require a distal pancreatectomy for extirpation:

  * total bilirubin <1.5 X institutional upper limit of normal*
  * AST(SGOT)/ALT(SGPT) <2 X institutional upper limit of normal*
  * creatinine <1.5X institutional upper limit of normal

    * Liver abnormalities in this range are consistent with pancreas cancer destruction from the tumor.
* The effects of MVT-5873 (HuMab-5B1) on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for 3 months after completion of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Subjects must agree to co-enrollment on the tissue collection protocol 13C0176, Tumor, Normal Tissue and Specimens from Patients Undergoing Evaluation or Surgical Resection of Solid Tumors.

EXCLUSION CRITERIA:

* Presence of disease outside the confines of a standard operation for subjects with periampullary cancers (pancreatic and cholangiocarcinoma).
* Presence of disease outside the liver for subjects with intrahepatic/hilar cholangiocarcinoma or metastatic colorectal cancer, other than a primary tumor for subjects with metastatic colorectal cancer.
* Subjects who are receiving any other investigational agents.
* Fewer than 28 days (or 5 half-lives for systemic agents, whichever is shorter) from the last day of prior anticancer therapy, including chemotherapy, hormonal, investigational, and or biological therapies and irradiation.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study

requirements.

-Active concurrent malignancies within the last five years other than the primary tumor

in subjects with metastatic colorectal cancer, basal or squamous cell skin carcinoma or non- medullary thyroid carcinoma.

* Pregnant women are excluded from this study because of the potential for teratogenic or abortifacient effects of the MVT-5873. Because there is an unknown but potential
* Subjects with active, Hepatitis B or C infection because of the potential for increased liver toxicity given the damaging effects of the virus.
* Allergic to chimeric, humanized or human antibodies.
* Received live vaccine within 4 weeks prior to first date of study intervention.
* Infection requiring hospitalization or herpes zoster treatment within 2 weeks prior to the first date of study intervention.
* Long-term infectious diseases (tuberculosis, fungal infections) active within 2 years prior to the first date of study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M Hernandez, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data is available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Derived] Gupta S, McDonald JD, Ayabe RI, Khan TM, Gamble LA, Sinha S, Hannah C, Blakely AM, Davis JL, Hernandez JM. Targeting CA 19-9 with a humanized monoclonal antibody at the time of surgery may decrease recurrence rates for patients undergoing resections for pancreatic cancer, cholangiocarcinoma and metastatic colorectal cancer. J Gastrointest Oncol. 2020 Apr;11(2):231-235. doi: 10.21037/jgo.2020.02.01. PMID 32399263
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-C-0039.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 - Pre-operative Escalation Doses of MVT-5873 (HuMab-5B1): Pre-operative escalation doses of MVT-5873, pancreatectomy or hepatectomy and post-operative MVT-5873 treatment
  MVT-5873: 1 mg/kg for pre-operative dose, 1 mg/kg during post-operative period
  pancreatectomy or hepatectomy: Pancreatectomy or hepatectomy
  Participants having low elevated liver function tests (LFTs), enrolled into pre-operative MVT-5873 escalation dose levels.
- Cohort 2 - Pre-operative Recommended Dose (RD) of MVT-5873 (HuMab-5B1): Pre-operative RD of MVT-5873, pancreatectomy or hepatectomy and post-operative MVT-5873 treatment
  MVT-5873: 1 mg/kg for pre-operative dose, 1 mg/kg during post-operative period
  pancreatectomy or hepatectomy: Pancreatectomy or hepatectomy
  Participants having moderate elevated liver function tests (LFTs), enrolled into pre-operative MVT-5873 escalation dose levels.
- Enrolled But Not Treated: Enrolled But Not Treated
Period: Overall Study
Arm/Group | Cohort 1 - Pre-operative Escalation Doses of MVT-5873 (HuMab-5B1) | Cohort 2 - Pre-operative Recommended Dose (RD) of MVT-5873 (HuMab-5B1) | Enrolled But Not Treated
Started | 8 | 1 | 1
Completed | 5 | 0 | 0
Not Completed | 3 | 1 | 1
Not completed — Screen failure | 0 | 0 | 1
Not completed — Ineligible | 1 | 0 | 0
Not completed — Physician Decision | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: One participant was enrolled but not treated. However, collected baseline data is reported here.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Pre-operative Escalation Doses of MVT-5873 (HuMab-5B1) | Cohort 2 - Pre-operative Recommended Dose (RD) of MVT-5873 (HuMab-5B1) | Enrolled But Not Treated | Total
Number analyzed (Participants) | 8 | 1 | 1 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 0 | 1 | 7
  >=65 years | 2 | 1 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.75 (6.39) | 69.7 (0) | 48.8 (0) | 63.65 (7.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 0 | 4
  Male | 5 | 0 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 3
  Not Hispanic or Latino | 6 | 1 | 0 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 0 | 3
  White | 5 | 1 | 0 | 6
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 1 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Disease Recurrence At 1 Year
Description: Disease recurrence is defined as new disease measurable on computed tomography (CT)/magnetic resonance imaging (MRI) that was not present on the baseline CT/MRI.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Pre-operative Escalation Doses of MVT-5873 (HuMab-5B1) | Cohort 2 - Pre-operative Recommended Dose (RD) of MVT-5873 (HuMab-5B1)
Number analyzed (Participants) | 8 | 1
Participants | 2 | 0

2. Primary Outcome: Number of Grade 3-5 Adverse Events Related and/or Not Related to Drug
Description: Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death related to adverse events.
Time Frame: Date treatment consent signed to date off study, approximately 29 months and 11 days, and 22 months and 21 days for cohort 1 and cohort 2 respectively.
Measure: Number; unit: Adverse events
Arm/Group | Cohort 1 - Pre-operative Escalation Doses of MVT-5873 (HuMab-5B1) | Cohort 2 - Pre-operative Recommended Dose (RD) of MVT-5873 (HuMab-5B1)
Number analyzed (Participants) | 8 | 1
Adverse events
  Grade 3 Abdominal pain - Not Related | 2 | 1
  Grade 3 Abdominal infection - Not Related | 1 | 0
  Grade 3 Alanine aminotransferase increased - Not Related | 2 | 1
  Grade 3 Alkaline phosphatase increased - Not Related | 0 | 1
  Grade 3 Anemia - Not Related | 5 | 1
  Grade 3 Aspartate aminotransferase increased - Not Related | 3 | 1
  Grade 3 Back pain - Not Related | 2 | 0
  Grade 3 Blood bilirubin increased - Not Related | 1 | 0
  Grade 3 Confusion - Not Related | 0 | 1
  Grade 3 Dyspnea - Not Related | 0 | 1
  Grade 3 Hematuria - Not Related | 1 | 0
  Grade 3 Hepatobiliary disorders- Other, Bile duct perforation - Not Related | 0 | 1
  Grade 3 Hyperglycemia - Not Related | 2 | 0
  Grade 3 Hypermagnesemia - Not Related | 1 | 0
  Grade 3 Hypertension - Not Related | 5 | 0
  Grade 3 Hypoalbuminemia - Not Related | 3 | 0
  Grade 3 Hypokalemia - Not Related | 3 | 0
  Grade 3 Hyponatremia - Not Related | 1 | 0
  Grade 3 Hypotension - Not Related | 1 | 0
  Grade 3 Lymphocyte count decreased - Not Related | 4 | 0
  Grade 3 Pharyngitis - Not Related | 1 | 0
  Grade 3 Thromboembolic event - Not Related | 1 | 0
  Grade 3 Urine output decreased - Not Related | 0 | 1
  Grade 3 Vomiting - Not Related | 0 | 1
  Grade 3 Alkaline phosphatase increased - Related | 2 | 4
  Grade 3 Anemia - Related | 3 | 3
  Grade 3 Aspartate aminotransferase increased - Related | 6 | 1
  Grade 3 Alanine aminotransferase increased - Related | 3 | 1
  Grade 3 Blood bilirubin increased - Related | 1 | 1
  Grade 3 Lymphocyte count decreased - Related | 0 | 1
  Grade 4 Aspartate aminotransferase increased - Not Related | 1 | 0
  Grade 4 Lymphocyte count increased - Not Related | 1 | 0
  Grade 4 Alkaline phosphatase increased - Related | 0 | 1
  Grade 5 Adverse Event - Not Related | 0 | 0
  Grade 5 Adverse Event - Related | 0 | 0

3. Secondary Outcome: Define Disease Free Survival (DFS) for Participants Treated With Preoperative MVT-5873
Description: Disease free survival is defined as resection day of surgery Day 0 (D0) until the time of documented clinical recurrence (radiographically or pathologically). In the absence of a knowable time of recurrence, time of death will be used as a surrogate. Clinical recurrence is cancer that has recurred during which the cancer could not be detected. This is judged on computed tomography (CT) or magnetic resonance imaging (MRI) as compared to the scan obtained after surgery and completion of the study drug.
Time Frame: An average of 15.17 months
Population: 5/8 participants were analyzed in cohort 1 because 2 participants were found to have peritoneal metastases on Day 0 and were taken off study, and 1 participant was taken off study due to study closure.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1 - Pre-operative Escalation Doses of MVT-5873 (HuMab-5B1) | Cohort 2 - Pre-operative Recommended Dose (RD) of MVT-5873 (HuMab-5B1)
Number analyzed (Participants) | 5 | 1
months | 14.5 [1 to 28] | 22 [NA to NA] — Full range cannot be calculated because the participant was taken off study due to study closure.

4. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Pre-operative Escalation Doses of MVT-5873 (HuMab-5B1) | Cohort 2 - Pre-operative Recommended Dose (RD) of MVT-5873 (HuMab-5B1)
Number analyzed (Participants) | 8 | 1
Participants | 7 | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 29 months and 11 days, and 22 months and 21 days for cohort 1 and cohort 2 respectively.
Arm/Group | Cohort 1 - Pre-operative Escalation Doses of MVT-5873 (HuMab-5B1) | Cohort 2 - Pre-operative Recommended Dose (RD) of MVT-5873 (HuMab-5B1)
All-Cause Mortality (participants affected / at risk) | 1/8 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/8 | 1/1
Other Adverse Events (participants affected / at risk) | 7/8 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Pre-operative Escalation Doses of MVT-5873 (HuMab-5B1) (N=8) | Cohort 2 - Pre-operative Recommended Dose (RD) of MVT-5873 (HuMab-5B1) (N=1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other, Bile duct perforation (Hepatobiliary disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Pre-operative Escalation Doses of MVT-5873 (HuMab-5B1) (N=8) | Cohort 2 - Pre-operative Recommended Dose (RD) of MVT-5873 (HuMab-5B1) (N=1)
Abdominal infection (Infections and infestations) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (6) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 6 (16) | 1 (5)
Alkaline phosphatase increased (Investigations) | 4 (11) | 1 (10)
Anemia (Blood and lymphatic system disorders) | 6 (24) | 1 (11)
Aspartate aminotransferase increased (Investigations) | 5 (21) | 1 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 3 (5) | 1 (2)
Chills (General disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 4 (17) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (14) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hypotension (Vascular disorders) | 2 (4) | 1 (1)
Lymph leakage (Vascular disorders) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (13) | 1 (4)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Thrush (Infections and infestations) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urine output decreased (Renal and urinary disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
White blood cell decreased (Investigations) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT03801915/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/15/NCT03801915/ICF_001.pdf